CLINICAL TRIAL: NCT07116356
Title: Molecular Characterization of Carbapenemase-Producing Enterobacterales Isolated From Clinical Samples in Egypt
Brief Title: Molecular Characterization of Carbapenemase-Producing Enterobacterales
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, assistant professor, Sohag University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: Soh-Mmed-25-7-10PD
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Carbapenem; enterobacterials,; Antibitic sensitivity; PCR
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Patients with enterobacterials infections (Experimental)
  Interventions: Diagnostic Test: Antibiotic administration; Diagnostic Test: Molecular detection of antibiotic resistance
- Group 2 patients with other bacterial infections (Experimental)
  Interventions: Diagnostic Test: Antibiotic administration; Diagnostic Test: Molecular detection of antibiotic resistance

INTERVENTIONS:
Diagnostic Test: Antibiotic administration — different samples were collected from patients admitted at oncology center at sohag
Diagnostic Test: Molecular detection of antibiotic resistance — Molecular detection of carbapenem resistant genes:
  * Extraction of nucleic acid from isolated organisms by boiling.
  * Primers will be used for detection of carbaenem resistant genes

SUMMARY:
Bacterial infections with carbapenem resistant pathogens are one of the major threats in immunocompromised patients, especially among cancer patients .Furthermore, Gram negative pathogens are becoming increasingly prevalent and have become an ongoing global health concern .Emergence of Gram-negative pathogens, especially Enterobacterales that avert many of the human defense mechanisms are alarmingly increasing and most of these pathogens are resistant to many of the in-use antibiotics including carbapenems .

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Sohag Oncology Center have different infections and isolated organism one of carbapenem resistant enterobacterales detected by antibiotic sensitivity test.

Exclusion Criteria:

* All patients admitted to Sohag Oncology Center having infections in different sites and isolated organisms are not one of enterobacterales and not carbapenem resistant.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Isolation of causative organism | 6 months

SECONDARY OUTCOMES:
Antibitic sensitivity test: | 2 months
Molecular detection of carbapenem resistant genes: | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://dx.doi.org/10.4103/ecdt.ecdt_40_23